CLINICAL TRIAL: NCT06141356
Title: [18F]Florbetazine ([18F]92) for Beta Amyloid PET Imaging in Alzheimer's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZineAD
Record Dates: First submitted 2023-11-11; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy participants: Drug: [18F]Florbetazine ([18F]92). A dosage of 10 mCi +/- 20% of Florbetazine will be injected by a PET-certified medical professional followed by 5ml 0.9% sodium chloride (normal saline) flush.
  Drug: [11C]PIB. A dosage range between 6.0-20.0 mCi of PIB will be injected by a PET-certified medical professional followed by 5ml 0.9% sodium chloride (normal saline) flush.
  Interventions: Drug: [18F]Florbetazine ([18F]92); Drug: [11C]PIB
- Patients with cognitive impairment: Drug: [18F]Florbetazine ([18F]92). A dosage of 10 mCi +/- 20% of Florbetazine will be injected by a PET-certified medical professional followed by 5ml 0.9% sodium chloride (normal saline) flush.
  Drug: [11C]PIB. A dosage range between 6.0-20.0 mCi of PIB will be injected by a PET-certified medical professional followed by 5ml 0.9% sodium chloride (normal saline) flush.
  Interventions: Drug: [18F]Florbetazine ([18F]92); Drug: [11C]PIB

INTERVENTIONS:
Drug: [18F]Florbetazine ([18F]92) — Participants will receive a single intravenous bolus injection of 10 mCi ± 20% of the investigational radiotracer [18F]Florbetazine and will undergo a PET/CT scan.
Drug: [11C]PIB — Participants will receive a single intravenous bolus injection of 6.0-20.0mCi of the investigational radiotracer [11C]PIB and will undergo a PET/CT scan.

SUMMARY:
[18F]Florbetazine ([18F]92) is a molecularly targeted imaging agent for Aβ protein with a novel diaryl-azine scaffold. It has shown specific binding affinity to Aβ aggregates in postmortem human AD brains and excellent brain pharmacokinetic properties with little non-specific retention in white matter in animal studies and a limited number of patients with Alzheimer's Disease (AD).

The purpose of the current study is to examine the binding properties of [18F]Florbetazine in human subjects and to compare the cortical and white matter binding with [11C]PiB or [18F]Florbetapir in the same subjects.

Imaging of the brain will be completed in healthy adult normal control participants and participants with cognitive impairment (including probable AD and dementia due to other conditions) to characterize [18F]Florbetazine uptake in the brain and its binding properties. [11C]PIB or [18F]Florbetapir PET imaging along with MRI will be completed in the same participants and the data will be compared with 18F-[18F]Florbetazine.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age ≥ 40 years
* Healthy participants or patients with probable Alzheimer's disease or with dementia due to other causes

Exclusion Criteria:

* Has allergy to [18F]Florbetazine or any of its excipients ;
* Has hypersensitivity to [11C]PIB or any of its excipients ;
* Incapable of providing written informed consent or lacking a legally authorized representative (LAR) to provide informed consent ;
* Unwilling or unable to undergo PET scans tracer injections ;
* Unwilling or unable to undergo MRI;
* Any condition that, in the Investigator's opinion, could increase the risk to the participant, limit the participant's ability to tolerate the research procedures, or interfere with the collection/analysis of the data (e.g., renal or liver failure, advanced cancer);
* Women who are currently pregnant or breastfeeding;

Ages: 40 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy participants of patients with probable Alzheimer's disease or with dementia due to other causes
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The non-displacable binding potential (BPND) of [18F]Florbetazine in healthy participants and patients with probable AD | 1 year
  Dynamic PET data in list-mode is required over 90 minutes in participants. The PET data will be reconstructed into specific dynamic series for kinetic modeling. The non-displacable binding potential (BPND) will be determined in target and reference tissues and compared between healthy participants and patients with probable AD.
The distribution volume ratio (DVR) of [18F]Florbetazine in healthy participants and patients with probable AD | 1 year
  Dynamic PET data in list-mode is required over 90 minutes in participants. The PET data will be reconstructed into specific dynamic series for kinetic modeling. The distribution volume ratio (DVR) will be determined in target and reference tissues and compared between healthy participants and patients with probable AD.
Comparison of the cortical and white matter binding of [18F]Florbetazine ([18F]92) with [11C]PIB in healthy participants and patients with cognitive decline | 2 years
  [18F]Florbetazine ([18F]92) PET and [11C]PIB PET will be conducted in the same subjects. standardized uptake value ratios of determined cortical and white matter regions will be calculated for both tracers and then compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, Peking Union Medical College Hopital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu M, Li Y, Liang M, Mao C, Dong L, Ge Q, Wu R, Ren C, Zhang H, Huang Z, Xing H, Yang X, Wang Y, Feng F, Cui M, Gao J, Huo L. The diagnostic performance of [18F]Florbetazine in Alzheimer's disease: a head-to-head comparison to [11C]PiB and [18F]Florbetapir. Eur J Nucl Med Mol Imaging. 2025 Aug;52(10):3557-3566. doi: 10.1007/s00259-025-07233-y. Epub 2025 Apr 4. PMID 40183954